CLINICAL TRIAL: NCT04002960
Title: Desaturation Validation of INVSENSOR00036
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TP-19901
Record Dates: First submitted 2019-06-27; First posted 2019-07-01 (Actual); Results first posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- INVSENSOR00036 (Experimental): All subjects who are enrolled into the test group and participate in data collection receive the noninvasive INVSENSOR00036 sensor
  Interventions: Device: INVSENSOR00036

INTERVENTIONS:
Device: INVSENSOR00036 — Noninvasive regional oximeter

SUMMARY:
This study is designed to evaluate the trending accuracy of a noninvasive regional oximetry measurement of somatic oxygen saturation. One investigational sensor (INVSENSOR00036) will be placed on the somatic site of the volunteer. The values obtained by the test sensor will be compared to the reference value obtained from an FDA-cleared sensor placed on the somatic site on the contralateral side.

ELIGIBILITY:
Inclusion Criteria:

* Subject is between 18 and 50 years of age.
* Subject weighs a minimum of 110 lbs and no more than 250 lbs unless subject is over 6 feet tall.
* Must have a hemoglobin value greater than or equal to 11 g/dL.
* Baseline heart rate ≥ 45 bpm and ≤ 85 bpm.
* Blood Pressure (Systolic BP < 140 mmHg and Diastolic BP < 90 mmHg).
* Carbon monoxide (CO) value less than or equal to 2.0% fractional carboxyhemoglobin (FCOHb)
* Subject has a physical status of ASA I or II (American Society of Anesthesiology Class I; Healthy subjects without any systemic disease at all. American Society of Anesthesiology Class II; subjects with mild systemic disease) as it applies to the systemic disease portion of the classification.
* Subject is able to read and communicate in English and understands the study and risks involved.

Exclusion Criteria:

* Subject is pregnant.
* Subject smokes (including e-cigarette use).
* Subject has a BMI > 35 and has been classified as morbidly obese or at an increased risk for participation by a medical professional.
* Subject has a history of fainting (vasovagal), blacking out or losing consciousness during or after a blood draw, or has a fear of blood draws.
* Subject has open wounds, inflamed tattoos or piercings and/or visible healing wounds that a medical professional renders them at an increased risk for participation.*
* Subject experiences frequent or severe headaches and/or migraine headaches, migraine auras, altitude sickness, and/or headaches accompanied by visual changes or sensitivity to light or sound.
* Subject has known drug or alcohol abuse and/or uses recreational drugs.
* Subject has experienced a concussion or head injury with loss of consciousness within the last year.
* Subject has any chronic bleeding disorders (i.e. hemophilia).
* Subject has any history of a stroke, myocardial infarction, seizures or heart attack.
* Subject has any cancer or history of cancer (not including skin cancer)*.
* Subject has a known neurological and/or psychiatric disorder (i.e. schizophrenia, bipolar disorder, Multiple Sclerosis, Huntington's disease) that interferes with the subjects' level of consciousness.
* Subject has any cardiac dysrhythmia(s) (i.e. atrial fibrillation) and has not received clearance by their physician to participate.
* Subject has Wolff-Parkinson-White Syndrome or Stokes-Adams Syndrome.
* Subject has taken anticoagulant medication within the last 30 days (excluding nonsteroidal anti-inflammatory drugs (NSAIDS)).
* Subject has donated blood within the past 4 weeks.
* Subject has taken opioid pain medication within 24 hours before the study.
* Subject has any type of infectious disease (i.e. Hepatitis, HIV, Tuberculosis, Flu, Malaria, Measles, etc.).
* Subject is taking medications known to treat any type of infectious disease.
* Subject has either signs or history of peripheral ischemia or carpal tunnel syndrome.
* Subject has had invasive surgery within the past year- including but not limited to major dental surgery*, appendix*, plastic surgery*.
* Subject has had invasive surgery within the past year- including but not limited gallbladder, major fracture repairs (involving plates/ screws), jaw surgery, urinary tract surgery, major ENT surgery, joint replacement or gynecological surgeries, heart surgery or thoracic surgery.
* Subject has symptoms of congestion, head colds, flu or other illnesses.
* Subject is claustrophobic and/or has generalized anxiety disorder.
* Subject has been in severe car accident(s) or a similar type of accident(s) requiring hospitalization within the last 12 months.
* Subject has chronic unresolved asthma, lung disease or respiratory disease.
* Subject is allergic to lidocaine, latex, adhesives, or plastic.
* Subject has a heart condition, insulin-dependent diabetes or uncontrolled hypertension.
* Subject has delivered vaginally, has had a pregnancy terminated, a miscarriage with hospitalization or had a C-section within the last 6 months.
* Subject has any medical condition which in the judgment of the investigator and/or medical staff, renders them ineligible for participation in this study (Discretion of investigator/study staff).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2019-07-05 (Actual); Study Completion 2019-07-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Masimo Corporation, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | INVSENSOR00036
Started | 23
Completed | 21
Not Completed | 2
Not completed — Withdrawn prior to Completion | 2

BASELINE CHARACTERISTICS:
Arm/Group | INVSENSOR00036
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 6
  Hispanic | 6
  Asian or Pacific Islander | 3
  Native American | 0
  Black or African American | 6
  Other | 0

OUTCOME MEASURES:

1. Primary Outcome: Trending Accuracy of INVSENSOR00036
Description: This study will evaluate the trending accuracy of the INVSENSOR00036 relative to the reference value obtained from the comparative FDA-cleared device.
Time Frame: 1-5 hours
Measure: Number; unit: percentage of regional oxygen saturation
Arm/Group | INVSENSOR00036
Number analyzed (Participants) | 21
percentage of regional oxygen saturation | 1.8

ADVERSE EVENTS:
Time Frame: 1 to 5 hours
Arm/Group | INVSENSOR00036
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 1/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | INVSENSOR00036 (N=23)
Chest tightness (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-09): https://cdn.clinicaltrials.gov/large-docs/60/NCT04002960/Prot_SAP_000.pdf